CLINICAL TRIAL: NCT05782621
Title: Acupoint Focused Ultrasound Versus Laserpuncture In Chronic Mechanical Neck Pain
Brief Title: Acupoint Focused Ultrasound Versus Laserpuncture In Mechanical Neck Pain
Acronym: MNP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Dina Ahmed Ahmed Asr, principle investigator Dina Ahmed Ahmed Asr, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004126
Record Dates: First submitted 2023-03-11; First posted 2023-03-23 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Neck Pain
Keywords: Acupoint Focused Ultrasound; Laserpuncture; Chronic Mechanical Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Intervention Model Description: Acupoint Focused Ultrasound and Laserpuncture
Who Masked: Investigator, Outcomes Assessor
Masking Description: opaque sealed envelop
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Acupoint focused ultrasound (Experimental): the patients will receive Acupoint focused ultrasound therapy three times a week for four weeks
  Interventions: Other: Acupoint focused ultrasound; Other: conventional treatment
- Laserpuncture (Experimental): the patients will receive Laserpuncture therapy three times a week for four weeks
  Interventions: Other: Laserpuncture; Other: conventional treatment
- conventional treatment (Active Comparator): the patients will receive conventional treatment three times a week for four weeks
  Interventions: Other: conventional treatment

INTERVENTIONS:
Other: Acupoint focused ultrasound — An ultrasound beam is normally pulsed in the ratio of 1:5. For perfect transmission of power from the treatment head to the body, the head will be applied perpendicularly to the skin surface. A stationary technique pulsed ultrasound (1 w/cm2) will be used. The application will be two minutes for each acupuncture point and the head will be glided to the next point in the same side; then to the other side for no more than 10 points, then the device will be turned off
  Arms: Acupoint focused ultrasound
Other: Laserpuncture — The laser tip (0.03 cm2 of beam area) will be positioned with the "probe" head directly on the acupuncture point, in a perpendicular position and in direct contact with the skin, and every point will be treated for 2 min, totaling 16 min of treatment, plus 4 min of rest, to standardize with the traditional acupuncture time, which is 20 min
  Arms: Laserpuncture
Other: conventional treatment — the patients will receive selective neck strengthening ex for (extension, flexion, sidebending, lateral rotation) and selective neck stretching ex for (extension, flexion, sidebending, lateral rotation)

SUMMARY:
this study will be conducted to compare the effect of Acupoint focused ultrasound and Laser puncture on pain intensity level, neck range of motion, and neck function in patient with chronic mechanical neck pain

DETAILED DESCRIPTION:
Neck pain is a musculoskeletal condition with a high prevalence that may affect the physical, social, and psychological aspects of the individual, contributing to the increase in costs in society and business. Neck pain was significantly associated with repetitive movement, activities that require lifting and moving loads, and being in sitting and leaning positions.Non specific neck pain is a multifactorial and very common condition in adult individuals, traditional acupuncture (TA) and laser puncture (LP) may be treatment options for certain individuals in such a condition. The laser will be placed at the specific acupuncture points: Tianzhu, Fengchi, Jianjing, and Jianzhongshu . Because ultrasound can deliver vibration energy to soft tissues noninvasively, ultrasound has been applied to diagnostic imaging and therapeutic applications. To use ultrasound for acupoint stimulation, a stimulation device was developed using focused ultrasound. The application of an ultrasound stimulus to the acupuncture meridian system has been found safe and effective in many common clinical entities. The Sonicator head is applied to the chosen location as in standard ultrasound therapy, with a gentle circular motion. forty five patients will be assigned randomly to three groups; experimental group 1 will receive acupoint focused ultrasound, experimental group 2 will receive laserpuncture and the control group will receive conventional treatment three times a week for four weeks.

ELIGIBILITY:
Inclusion Criteria:

All subjects will be referred by the orthopedist. Cervical pain is episodic chronic, having occurred and recurred over regular or irregular intervals of time over at least the last 3 months.

The subject is willing and able to refrain from non-study procedure therapies for the management of neck pain throughout study participation.

Age ranged from 30-60 years BMI ranged from (25-30kg/m2)

Exclusion Criteria:

Cervical pain is undiagnosed or has been diagnosed as being other than of benign musculoskeletal origin.

Tension myositis syndrome. Osteoporosis with compression fractures. Congenital deformity of spine. Current active chronic pain disease. Cancer or cancer treatment in the past 6 months. Use of the following analgesics within 7 days of study onset - paracetamol, acetominophen, non-steroidal anti-inflammatory drugs (NSAIDs), compound analgesics, topical analgesics.

Use of the following muscle relaxants within the prior 30 days of study onset - cyclobenzaprine, diazepam, meprobamate.

Ages: 30 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2023-03-30 (Estimated); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
pain intensity | up to four weeks
  pain will be measured by visual analogue scale. It is a vertical or horizontal 100 mm line graduated by different levels of pain, starting from 0 (no pain) till 100 (worst pain)
Disability | up to four weeks
  The Copenhagen Neck Functional Disability Scale will be used to evaluate the disability experienced by patients with neck pain. it consists of 15 items. These items are individually answered by either 'yes', 'occasionally' or 'no'. For questions one till five, a 'yes' indicates a good function. For questions six till fifteen, a 'no' indicates a good function. A good function receives a score of zero, a poor function receives a score of two and the answer 'occasionally' always receives a score of one. Afterwards, we add up all the scores of the questions to form the total score. This total score ranges from 0 to 30.The total score determines the level of functional disability, in which higher numbers represent a higher level of disability. A score of 0 indicates that there are no neck complaints present whereas 30 indicates that the patient is extremely disabled as a result of the neck complaints

SECONDARY OUTCOMES:
cervical range of motion | up to four weeks
  The digital goniometer will be used for measuring cervical range of motion